CLINICAL TRIAL: NCT01051427
Title: Control of Epistaxis With Surgiflo
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Now we use better procedures for the patient instead of nasal catheter for epistaxis. So it would be unethical to use the nasal catheter to complete the trial.
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, Gonzalo de los Santos, MD, PhD, Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ORLEPI1; ORLEPI1 (Other: Ethical Committee of the Ramon y Cajal hospital)
Record Dates: First submitted 2010-01-14; First posted 2010-01-18 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Epistaxis
Keywords: Nasal packing; Haemostatic matrix; Epistaxis control
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nasal catheter (Active Comparator): In this arm will be the patients with epistaxis that cannot be stopped with anterior nasal packing and are randomized not to put Surgiflo. So they receive the usual treatment with a nasal catheter balloon into the nose.
  Interventions: Device: Nasal catheter
- Surgiflo (Experimental): In this arm will be the patients with epistaxis that cannot be stopped with anterior nasal packing and are randomized to put into the nose Surgiflo.
  Interventions: Device: Surgiflo

INTERVENTIONS:
Device: Surgiflo — Before to put a nasal catheter to stop nasal bleeding when anterior packing fails, we'll try to stop bleeding with Surgiflo.
  Other Names: Surgiflo haemostatic matrix.
  Arms: Surgiflo
Device: Nasal catheter — In patients randomized not to put Surgiflo, we use a nasal catheter to try to stop nasal bleeding.
  Other Names: Invotec, Ultra Stat, nasal catheter.
  Arms: Nasal catheter

SUMMARY:
This is a blind trial to test if Surgiflo is effective in posterior epistaxis. After the investigators see than anterior tamponade is not effective stopping epistaxis, the investigators try using Surgiflo and if it does not work the investigators continue with a nasal catheter. This is the usual way to stop nasal bleeding, but is painful and has serious after-effects in the nose. Surgiflo is a hemostatic matrix that can be put into the nose, painlessly and easily. So the investigators think it can be useful controlling nasal bleeding, so the investigators could avoid to put nasal catheters in these patients.

DETAILED DESCRIPTION:
Epistaxis is one of the most frequent diseases in Otolaryngology emergencies. Most of them are anterior and stop with an anterior packing. Some of them does not stop with this, therefore the investigators have to put into the nose a catheter balloon. This is very painful and has many after-effects in the nose.

Surgiflo is a haemostatic matrix used for bleeding.

The investigators have design a trial to know if some people can benefit from Surgiflo instead to put a nasal catheter.

This a randomized trial with two arms. In one arm the investigators will put surgiflo and not in the other.The patient will be admitted to the hospital. The investigators will see the difference in the hospital staying and in the effects in the nose, including discomfort or pain. The investigators will report age, gender, other diseases or treatments of the patients,type and length of bleeding, transfusions needed, arterial tension, coagulation. To do that the investigators will make hematological tests for haemoglobin and coagulation. To know the discomfort of the device the investigators will give the patient an analog visual scale in the moment the investigators will put the device, the day after and in any of the next visits. The patient can go home again after 16h without bleeding and the investigators will see the patient again in the office after 15 days, 1, 3 and 6 months.

All the patients will receive the same analgesic protocol so the investigators can compare the discomfort.

The investigators have make statistic analysis, and they will need 24 patients for this trial. The investigators will need 2 years, approximately, to recruit them.

ELIGIBILITY:
Inclusion Criteria:

* Patients with epistaxis in emergency room.
* Epistaxis does not stop with anterior nasal packing.

Exclusion Criteria:

* Pregnancy
* Allergy or intolerance to any component of Surgiflo.
* Septal perforation.
* Nasal surgery within 3 months previous to epistaxis.
* Patients admitted to hospital for other reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2010-03; Primary Completion 2012-03 (Estimated); Study Completion 2012-08 (Estimated)

PRIMARY OUTCOMES:
Days admitted to the hospital related to epistaxis | From intervention (nasal catheter or Surgiflo) until 1 day after discharge

SECONDARY OUTCOMES:
Discomfort and troubles related to the device used to treat epistaxis. | Within 6 months after tamponade

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo de los Santos, MD, PhD, Principal Investigator — Ramon y Cajal Hospital
Locations (1):
- Ramon y Cajal Hospital, Madrid, Madrid, Spain

REFERENCES:
- [Background] Mathiasen RA, Cruz RM. Prospective, randomized, controlled clinical trial of a novel matrix hemostatic sealant in patients with acute anterior epistaxis. Laryngoscope. 2005 May;115(5):899-902. doi: 10.1097/01.MLG.0000160528.50017.3C. PMID 15867662
- [Background] Chandra RK, Conley DB, Kern RC. The effect of FloSeal on mucosal healing after endoscopic sinus surgery: a comparison with thrombin-soaked gelatin foam. Am J Rhinol. 2003 Jan-Feb;17(1):51-5. PMID 12693656
- [Background] Woodworth BA, Chandra RK, LeBenger JD, Ilie B, Schlosser RJ. A gelatin-thrombin matrix for hemostasis after endoscopic sinus surgery. Am J Otolaryngol. 2009 Jan-Feb;30(1):49-53. doi: 10.1016/j.amjoto.2007.11.008. Epub 2008 Jun 16. PMID 19027513
- [Background] Gudziol V, Mewes T, Mann WJ. Rapid Rhino: A new pneumatic nasal tamponade for posterior epistaxis. Otolaryngol Head Neck Surg. 2005 Jan;132(1):152-5. doi: 10.1016/j.otohns.2004.04.005. PMID 15632931